CLINICAL TRIAL: NCT00615121
Title: Genetics of Peripheral Artery Disease
Brief Title: Genetics of Peripheral Artery Genomics
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00008270; 4814-07 (Other: Duke legacy protocol number)
Record Dates: First submitted 2008-02-03; First posted 2008-02-14 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Peripheral Artery Disease
Keywords: Smoking; Hypertension; Diabetes; Cardiovascular disease; Renal Failure
MeSH Terms: conditions — Peripheral Arterial Disease; Smoking; Hypertension; Diabetes Mellitus; Cardiovascular Diseases; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral artery samples collected from patients are stored in -80celcius refrigerator for future analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- arteries from PAD patients: peripheral arteries from patients undergoing amputation for end stage peripheral arterial occlusive disease
- arteries from Free Fib transfers: peripheral arteries from patients without evidence of peripheral arterial occlusive disease

SUMMARY:
Peripheral artery disease is a disease that contributes to significant morbidity and mortality of millions of Americans yearly. Very little is known about the pathophysiology of atherosclerosis in peripheral artery disease. We plan to collect peripheral arteries and muscle tissue from patients undergoing amputation for end stage peripheral arterial occlusive disease. By extracting the RNA from these arteries and tissues and comparing them with RNA expression from normal arteries, we hope to have a better understanding of the pathophysiology of atherosclerosis in this setting. We aim to prove the hypothesis that a novel gene expression pattern can be discovered by the successful extraction of RNA from plaques from human peripheral arteries.

DETAILED DESCRIPTION:
Patients scheduled to undergo lower extremity amputation will be consented for extraction of plaque from the carotid artery or arterial tissue from the amputated limbs. The surgeon will perform the amputation, then the harvest team will collect arterial tissue from amputated limbs. These samples will be immersed in RNALater solution to preserve the integrity of the RNA. Tissues will stored at -80oC in the RNALater until the RNA is later extracted using a standardized protocol. The RNA will be examined for quality using an Agilent bioanalyzer, and will then be processed on Affymetrix U133A chips for gene expression data. The data will be analyzed with the MATLAB software package.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing amputations for peripheral artery disease
* Patients undergoing free fibular transfer

Exclusion Criteria:

* those that are not able to consent to the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with peripheral artery occlusive disease.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2004-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Discover novel gene expression pattern in peripheral arterial disease | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Lawson, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States